CLINICAL TRIAL: NCT03128554
Title: Smoking Reduction: Testing a Novel Approach to Cessation in Primary Care Practice Settings: A Pilot Study
Brief Title: Smoking Reduction: Testing a Novel Approach to Cessation in Primary Care Practice Settings
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding was withdrawn in January 2020. Covid-19 pandemic prevented the study from continuing to a point where it would need to be restarted. Multiple participants dropped out throughout pandemic.
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: University of Ottawa (Other); The Ottawa Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 20170061-01H
Record Dates: First submitted 2017-04-12; First posted 2017-04-25 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Smoking Cessation
Keywords: Not Ready to Quit; Primary Care; Tobacco; Reduce to Quit; Smoking Reduction
MeSH Terms: conditions — Smoking Cessation; Smoking Reduction | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention with Training and Materials (Experimental): Clinics randomized to the intervention group will receive a one time, 2-hour Continuing Medical Education/Group Learning training session on the smoking reduction intervention model, along with provider and patient handouts.
  Interventions: Other: Intervention with Training and Materials
- Usual Care (No Intervention): Clinics randomized to the control group will not be exposed to the intervention program.

INTERVENTIONS:
Other: Intervention with Training and Materials — Peer-Led Continuing Medical Education Session and Provider/Patient Handouts
  Arms: Intervention with Training and Materials

SUMMARY:
Traditional models of smoking cessation focus on delivering advice and counseling to quit and providing assistance to patients ready to quit smoking, but do not actively intervene with patients who are not ready to quit (NRTQ). This abrupt cessation approach is often not an appealing option to those not ready to quit, however, a reduction approach can seem more attainable and engaging. In response to this need, this smoking cessation intervention has been developed.

This research is part of a pilot study to assess the feasibility of introducing a NRTQ intervention in a primary care setting. This study will also assess the effectiveness of increasing the number of smoking reduction interventions delivered, provider confidence and satisfaction, relative to control practice. Outcomes will be assessed by a pre-survey and a three-month follow-up survey, administered to all study participants. All study participants will also be asked to fill out brief NRTQ consult forms for each NRTQ patient they encounter for a two-week period. Additionally, participants randomized to the intervention arm will receive training, and access to tools and resources.

DETAILED DESCRIPTION:
3.0 HYPOTHESIS TO BE TESTED The intervention program will be feasible to introduce into primary care practices. The intervention program will also be effective in increasing the number of smoking reduction interventions delivered and provider confidence, relative to control practice. Providers in the intervention condition will be satisfied with the intervention and tools provided.

4.0 RELEVANCE TO THE ADVANCEMENT OF THE TREATMENT OF NICOTINE DEPENDENCE The Ministry of Health and Long Term care recently published an updated action plan on smoking cessation in Ontario (24). This action plan focuses on smoking prevention and cessation rather than harm reduction in smokers not ready to quit, which accounts for the majority of smokers in Ontario (24). Previous studies have demonstrated that smoking reduction strategies employing NRT can lead to smoking cessation in smokers not yet ready to quit (12). This pilot study aims to determine the feasibility of introducing a multi-component intervention program for primary care providers to target the unmotivated to quit smoker. If successful it will inform a larger trial throughout the OMSC platform to further evaluate the effectiveness of the smoking cessation through reduction approach. This might result in a shift in smoking cessation culture in Canada to include harm reduction as an approach to engage the smoker who is not ready to quit.

5.0 METHODS TO BE USED 5.1 Design A two-armed, cluster randomized controlled pilot study will be conducted. Primary care practices will be randomized to one of two study arms: the 'control' group or the 'intervention' group. Ten primary care practices will be randomly assigned to one of the two arms (5 practices per arm).

The study design schema and timeline for the collection of outcome data and intervention activities is presented in Appendix A -- Study Flow Diagram and Timeline.

5.2 Setting and Participants Ten primary care practices (5 per study arm) from the existing Ottawa Model for Smoking Cessation (OMSC) primary care network will be recruited from within the province of Ontario, over a 3-month recruitment period. We will recruit ≥ 40 Medical Doctors (MD), Nurse Practitioners (NP), Registered Nurses (RN), and pharmacists for participation.

5.3 Procedures 5.3.1 Recruitment of OMSC primary care practices A study invitation letter [Appendix C -- Study Invitation Letter] will be emailed to OMSC partner sites [Appendix B -- Participant Recruitment Email] located in the Champlain, South East, or Central East Local Health Integration Networks (LHINs), addressed to the lead physician, executive director or clinic manager. A member of the research team will place a follow-up phone call approximately one week later to inquire about the interest in study participation [Appendix D -- Telephone Script]. Once they have agreed to take part in the study, an email will be sent to all eligible providers within that clinic, asking them to take part in the study [Appendix E -- Provider Recruitment Email] with an attached invitation letter [Appendix F -- Study Invitation Letter for Providers]. All primary care providers from eligible participating practices will provide informed consent [Appendix G -- Telephone Script for Obtaining Verbal Consent].

Participants who wish to withdraw from the study after being consented must provide a letter to the PI [Appendix H -- Participant Withdrawal Letter].

If we are unable to recruit all ten primary care practices within the above-mentioned Local Health Integrated Networks (LHINs), we will expand recruitment to all LHINs within Ontario [Appendix Q-Eligible Sites for Expansion].

5.3.2 Allocation to treatment A two-armed, cluster randomized controlled pilot study will be conducted. Primary care practices will be randomized to one of two study arms: the 'control' group or the 'intervention' group. Randomization will be performed by the UOHI research methods group who will not be directly involved in the study. Primary care clinics will not be blind to the group assignment however the investigator responsible for statistical analysis will remain blinded to group assignment. The Ottawa Health Science Network Research Ethics Board (OHSN-REB) will approve this study.

5.3.3 Data Collection

5.3.3.1 Pre- and Post-Assessment Survey At baseline, participating primary care providers will complete a brief study questionnaire, which will document demographic characteristics of providers (age, gender, practice model, geographic location), provider knowledge and confidence in addressing smoking cessation with patients not ready to quit, and assess each provider's current practice with NRTQ patients. These surveys will be mailed to a contact person at the clinic, who will distribute and collect the surveys to return them to the Ottawa Model for Smoking Cessation [Appendix K -- Pre-Survey Instructions]. At the 3-month follow-up, providers will also complete a second survey which will re-assess provider confidence and satisfaction with the intervention program [Appendix I -- Pre and Post Provider Surveys]. These surveys will again be mailed out to a contact person at the clinic, who will distribute and collect the surveys to return to the Ottawa Model for Smoking Cessation [Appendix L -- Post-Survey Instructions].

5.3.3.2 Not Ready to Quit (NRTQ) Consult Form At the 3-month follow-up, providers will complete a brief consult form [Appendix J -- Tools and Resources] for a two week period which will document the number of smoking reduction interventions completed with NRTQ patients. The consult form will be provided to both the control and intervention groups, and a chart audit will assess the number of smoking reduction interventions provided. The consult forms will be mailed to a contact person at the clinic who will distribute and collect the packages of forms, and return them to the Ottawa Model for Smoking Cessation [Appendix M -- NRTQ Consult Form Instructions]. The packages will also contain a letter for providers with instructions on how to complete the forms, as well as a form indicating when they started and completed NRTQ Consult Forms [Appendix N -- NRTQ Provider Instruction].

5.3.4 Group Comparators 5.3.4.1 Intervention group The intervention program will focus on the sub-population of tobacco users who report they are not ready/motivated to quit smoking in the next 30 days but are willing to cut back on smoking over the next 3 months. All providers randomized to this group will receive a 2-hour Continuing Medical Education (CME)/Group Learning (GLS) training session on the smoking reduction intervention model. The CME/ GLS will be delivered by a peer primary care physician. To support delivery of the reduction program in primary care settings, providers in the intervention group will receive a not ready to quit (NRTQ) consult form, provider resource, and patient handout which may be integrated into EMR systems as appropriate. [Appendix J -- Tools and Resources]

5.3.4.2 Control group Clinics randomized to the control group will not be exposed to the intervention program. Providers in this group however receive the NRTQ consult form for data collection purposes [Appendix J -- Tools and Resources].

5.4 Outcome measures

5.4.1 Participation rate (i.e. Practitioner recruitment). The study will evaluate the number of providers who agree to participate divided by the total number of providers who are sent an invitation letter. By measuring participation rate, it will inform recruitment for a larger study.

5.4.2 NRTQ consult completion rate. The number of NRTQ consults completed per physician in the intervention group and the control group will be evaluated and compared. It is anticipated that providers that have received the intervention will have a higher NRTQ consult completion rate. This will also evaluate the uptake of the NRTQ consult form by health care providers.

5.4.3 The number of reduction interventions provided by providers. A chart audit of both the intervention and control groups will measure the number of reduction interventions provided in the NRTQ population. This will assess the feasibility of this intervention in primary care as well as act as a surrogate to inform a larger trial of the receptiveness patients have to a smoking intervention when they are NRTQ. A chart audit instruction sheet and documentation form will be faxed to a contact person at the clinic who will record the total number of NRTQ patients seen by each participating provider during their respective two-week period. The clinic contact person will return the form via fax to the Ottawa Model for Smoking Cessation [Appendix R - Number of Patients NRTQ].

5.4.4 Provider confidence in addressing tobacco use among patients NRTQ. Provider confidence will be measured in a pre and post intervention surveys completed by participating health care providers in both the intervention and control groups. This will evaluate if providing a 2-hour Continuing Medical Education (CME)/Group Learning (GLS) training session on the smoking reduction intervention model will alter provider confidence in intervening in the NRTQ population and help inform a larger study. If provider confidence is not affected by the NRTQ CME/GLS, the intervention will need to be re-evaluated prior to a larger study.

5.4.5 Provider satisfaction with the smoking reduction intervention program. Provider satisfaction with the smoking reduction intervention program will be assessed in the intervention group only. Summary statistics on provider satisfaction will help inform a larger study as well as identify if the intervention is acceptable for primary health care providers.

5.5 Sample size As this is a feasibility study, the sample size was dictated by available resources. We plan to recruit five sites per study arm, and a minimum of four providers per site, giving a minimum total of 40 health care providers from which to generate the estimates of intervention efficacy (defined as the number of reduction interventions performed, excluding dedicated smoking cessation visits and unscheduled visits).

5.6 Statistical analysis For the primary data analyses, we will compare the mean number of NRTQ consults between groups using a t-test that incorporates a variance inflation factor to account for the effect of clustering. If there are relevant baseline differences between groups, we will use Generalized Estimating Equations (GEE) to account for clustering and co-variates. Similar analytics will be applied for comparing confidence levels between the two groups. Summary statistics will be calculated for provider satisfaction with the intervention in the smoking reduction group.

5. 7 Potential problems and possible approaches for overcoming them There may be concerns about the feasibility of primary care practice and provider recruitment, the completion rate for the experimental intervention and loss-to-follow-up. Our research team has extensive experience conducting clinical trials of smoking cessation interventions (5, 6, 15). There are presently 31 eligible primary care practices in the Champlain, South East, and Central East LHINs [Appendix O -- Eligible Primary Care Practices], within the province of Ontario, which suggests we will be able to recruit the required sample size of ten primary care practices with relative ease.

5.8 Ethical issues relating to the involvement of human subjects Trial design and conduct has been informed by Good Clinical Practice (GCP), an international ethical and scientific quality standard for designing, conducting, recording and reporting trials that involve the participation of human subjects. Compliance with this standard provides public assurance that the rights, safety and well-being of trial subjects are protected, consistent with the principles that have their origin in the Declaration of Helsinki, and that the clinical trial data are credible. The final study protocol will be reviewed and approved by the Ottawa Health Science Network Research Ethics Board REB. The trial will be reported in accordance with CONSORT guidelines for cluster randomized trials (23), and will be registered with clinicaltrials.gov.

ELIGIBILITY:
Inclusion Criteria:

* Primary care practice from the existing OMSC network
* Primary care practice is staffed by ≥ 4 MDs/NPs/RNs/Pharmacists
* A minimum of four clinicians within the practice are willing to participate

Exclusion Criteria:

* Actively using a Reduce to Quit protocol in practice

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of Providing the Intervention Measured by the Participation Rate | 1 year
  The feasibility of introducing a not ready to quit (NRTQ) intervention in a primary care setting by measuring the participation rate (i.e. Practitioner recruitment). The study will evaluate the number of providers who agree to participate divided by the total number of providers who are sent an invitation letter.
Feasibility of Providing the Intervention Measured by the Consult Completion Rate | 1 year
  The feasibility of introducing a not ready to quit (NRTQ) intervention in a primary care setting by measuring the NRTQ consult completion rate. The number of NRTQ consults completed per physician in the intervention group and the control group will be evaluated and compared.

SECONDARY OUTCOMES:
Increasing the number of reduction interventions provided by providers | 3 months
  This outcome is measured by the completion of the NRTQ forms and a chart audit. The chart audit will determine how many not ready to quit patients were seen by the provider as compared to how many of those patient received a reduction intervention. A reduction intervention is tracked by the provider using the "Not Ready to Quit" consult form. The language "reduction" is important to keep in our study because the word "change" is not specific enough. We are measuring the amount of reduction smoking cessation interventions specifically - meaning gradual cessation as compared to abrupt cessation.
Increasing provider confidence in addressing tobacco use among patients NRTQ | 3 months
  Provider confidence will be measured in a pre and post intervention surveys completed by participating health care providers in both the intervention and control groups. This will evaluate if providing a 2-hour Continuing Medical Education(CME)/Group Learning (GLS) training session along with resources on the smoking reduction intervention model will alter provider confidence in intervening with the NRTQ population and help inform a larger study. Provider confidence is measured on a 10 point scale (1 being not very confident and 10 being extremely confident)
Assessing provider satisfaction with the smoking reduction intervention program: post-intervention survey | 3 months
  Provider satisfaction with the smoking reduction intervention program will be assessed in the intervention group only through a post-intervention survey. Provider satisfaction is based on the selection of one of three choices: "Not satisfied", "somewhat satisfied" or "very satisfied"

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Murley, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website for the Ottawa Model for Smoking Cessation — http://ottawamodel.ottawaheart.ca/